CLINICAL TRIAL: NCT04616378
Title: Design, Prototyping, and Testing of a Robotic Prosthetic Leg
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5200345
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Amputation; Traumatic, Leg, Lower

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 2 Prescribed Prosthesis (Other): Participants everyday use of prosthesis
  Interventions: Other: Phase 2 Prescribed Prosthesis
- Phase 2 Robotic Prosthetic Leg (Experimental): Robotic prosthetic leg with powered knee and passive ankle
  Interventions: Other: Phase 2 Robotic Prosthetic Leg
- Phase 3 Prescribed Prosthesis (Other): Participants everyday use of prosthesis
  Interventions: Other: Phase 3 Prescribed Prosthesis
- Phase 3 Robotic Prosthetic Leg (Experimental): Robotic prosthetic leg with powered knee and passive ankle
  Interventions: Other: Phase 3 Robotic Prosthetic Leg
- Phase 3 No Prosthesis (Experimental): Participant performs tasks with no prosthetic device attached
  Interventions: Other: Phase 3 No Prosthesis

INTERVENTIONS:
Other: Phase 2 Prescribed Prosthesis — Everyday used prosthesis that was prescribed by their physician.
  Arms: Phase 2 Prescribed Prosthesis
Other: Phase 2 Robotic Prosthetic Leg — The RPL consists of a passive-dynamic ankle, powered knee, and an on-board inertial measurement sensors with an on-board kinetic and kinematic data collection system for analysis.
  Arms: Phase 2 Robotic Prosthetic Leg
Other: Phase 3 No Prosthesis — No prosthetic device is attached.
  Arms: Phase 3 No Prosthesis
Other: Phase 3 Robotic Prosthetic Leg — The RPL consists of a passive-dynamic ankle, powered knee, and an on-board inertial measurement sensors with an on-board kinetic and kinematic data collection system for analysis.
  Arms: Phase 3 Robotic Prosthetic Leg
Other: Phase 3 Prescribed Prosthesis — Everyday used prosthesis that was prescribed by their physician.
  Arms: Phase 3 Prescribed Prosthesis

SUMMARY:
The purpose of this graduate student research study is to test that a specifically designed and novel robotic prosthetic leg (RPL) is feasible, safe and improves symmetry, efficiency, and metabolic function during sit-to-stand and stand-to-sit transitions as compared to the subject's prescribed device, and as compared to no device at all.

DETAILED DESCRIPTION:
Phase 2 case study

* Two subjects will be fitted with a heart rate monitor and with an adapted waist belt with mobile phone attached.
* RPL alignment will be verified.
* The subjects will use the RPL in parallel bars 10 times and take rests as needed in a chair.
* The subjects will perform the timed up and go test (TUGT), 10-meter walk test (10MWT), and the 6-minute walk test (6MWT).
* The subjects will be fitted with retro-reflective markers.
* The subjects will be fitted with a portable oxygen uptake analyzer.
* A 4D motion-capture camera system will be used while performing TUGT and five times sit to stand (5XSTS).
* The subjects will perform the above tests in their prescribed daily-wear prosthesis, and then in the RPL.
* The subjects will complete the activities-based balance confidence (ABC) scale test.
* The subjects will be asked a series of open-ended questions regarding the experience, while being audio recorded.

Phase 3 pilot study

* Twenty subjects will be randomized into three treatment arms (no prosthesis, prescribed prosthesis, RPL).
* The subject will be fitted with a heart rate monitor.
* The subject will be fitted with a portable oxygen uptake analyzer.
* The subject will be fitted with the RPL, and the alignment of the RPL will be confirmed before testing.
* The subject will be fitted with retro-reflective markers.
* A 4D motion-capture camera system and force-plate will be used while performing the 5XSTS test in the assigned randomized condition. The test will be performed three times in each condition.
* The subject will return two more times to complete the tests in the remaining randomized conditions, with a two-week washout period between sessions.
* The subject will be given the ABC scale test in the beginning and at the end of this study.
* The subject will complete the technology attitudes questionnaire (TAQ).
* In total, subject participation will last 1 hour per day, for three sessions, two weeks apart.

ELIGIBILITY:
Phase 2

Inclusion Criteria:

* unilateral limb-loss.
* amputation or knee disarticulation/transfemoral amputation
* can walk with a variable cadence (Level K3) or play sports (Level K4)
* uses a prosthesis for walking daily
* can stand for 30 seconds on one limb
* can follow one-step commands.

Exclusion Criteria:

* Those who can not walk with a variable cadence (Level K1 and K2)
* compromised skin on the residual limb (stump)
* uncontrolled swelling
* missing more than one limb

Phase 3

Inclusion Criteria:

* unilateral knee disarticulation or transfemoral amputation.
* can walk at a single speed (Level K2), can walk with a variable cadence (Level K3) or play sports (Level K4)
* can follow one step commands.

Exclusion Criteria:

* Those who do not use prosthesis for walking (Level K1)
* compromised skin on the residual limb (stump)
* uncontrolled swelling
* missing more than one limb

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | two weeks
  The participant sits in a standard armchair with any assistive device used for walking nearby. The participant stands and at a self-selected walking speed, walks 3 meters, turns, and walks back to the chair, and sits down. A stopwatch records the time to of the test (in seconds).

SECONDARY OUTCOMES:
10 meter walk test | one week
  The participant will be timed as he/she walks a known distance of 10 meters to determine his/her self-selected walking velocity (distance/time).

OTHER OUTCOMES:
6 minute walk test | one week
  This test measures distance walked in six minutes to assess the participant's physical endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Daher, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States